CLINICAL TRIAL: NCT06993805
Title: Evaluation of Our Practice Advisory (OPA) Interventions on Hemoglobin A1c (A1c) and Thyroid-Stimulating Hormone (TSH) Short Interval Ordering
Brief Title: Evaluating a Our Practice Advisory (OPA) to Optimize Hemoglobin A1c (A1c) and Thyroid-Stimulating Hormone (TSH) Test Orders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Catherine A. Sarkisian, Associate Professor of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB-25-0120
Record Dates: First submitted 2025-04-30; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Physician Workflow; Resource Utilization
Keywords: Clinical Decision Support; Laboratory Test Optimization; Resource Utilization; Our Practice Advisory (OPA)

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OPA Intervention Group (Experimental): Providers in this group will receive a Our Practice Advisory (OPA) through the electronic health record (EHR) system when ordering Hemoglobin A1c (A1c) and Thyroid-Stimulating Hormone (TSH) tests. The OPA will prompt providers to reconsider the test if it was ordered within the previous 30 days, aligning with evidence-based guidelines to reduce unnecessary testing.
  Interventions: Behavioral: OPA
- Control Group (No Intervention): Providers in this group will not receive a Our Practice Advisory (OPA) through the Electronic Health Record (EHR) system when ordering Hemoglobin A1c (A1c) and Thyroid-Stimulating Hormone (TSH) tests. This group represents the current standard of care, with no additional prompts or alerts implemented.

INTERVENTIONS:
Behavioral: OPA — The Our Practice Advisory (OPA) intervention is a behavioral nudge integrated into the electronic health record system. It is designed to prompt providers to reconsider ordering Hemoglobin A1c (A1c) and Thyroid-Stimulating Hormone (TSH) tests if a similar test was performed within the previous 30 days. The OPA aligns with evidence-based guidelines to reduce unnecessary testing, improve resource utilization, and optimize patient care by enhancing clinical decision-making at the point of order entry.
  Arms: OPA Intervention Group

SUMMARY:
Our Practice Advisory (OPA) are essential tools in clinical decision-making. The alerts are designed to guide providers towards evidence-based practices and improve patient outcomes. The focus of this initiative is on Hemoglobin A1c (A1c) and Thyroid-Stimulating Hormone (TSH) testing, with the goal of addressing unnecessary repeat testing within a 30-day timeframe, which rarely yields significant new insights. Although randomization occurs at the patient level, the primary outcome of this study focuses on provider behavior and decision-making.

By focusing on this specific intervention, the study aims to optimize resource use, align test ordering with evidence-based guidelines, and support improved patient outcomes. The results of this evaluation will help refine OPAs and guide broader strategies for implementing clinical decision support tools across healthcare systems.

DETAILED DESCRIPTION:
The purpose of this Quality Improvement (QI) initiative is to evaluate the impact of a randomized Our Practice Advisory (OPA) intervention on physician ordering behavior of Hemoglobin A1c (A1c) and Thyroid-Stimulating Hormone (TSH) tests within a 30-day interval from the prior test. The OPA will fire when an A1c or TSH are ordered within 30 days of a prior result (these short-interval tests are widely considered unnecessary) and will ask providers to reconsider the order. This study will evaluate the effectiveness of this intervention by randomizing patients 1:1 such that physicians caring for the patient will either (1) receive the OPA or (2) not receive the OPA if the providers order a short-interval test. This study is being conducted for a primary QI intent, as the results will (1) dictate if the short-interval OPA should be implemented across all patients, and (2) if this short-interval OPA should be applied to other labs aside from A1c and TSH. In these ways, the purpose of this study is to directly inform health system operations.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Inpatient or observation stays within UCLA Health System hospitals
* Hemoglobin A1c (A1c) and Thyroid-Stimulating Hormone (TSH) ordered, AND this lab was ordered and resulted within the prior 30 days

Exclusion Criteria:

* Have an A1c or TSH ordered and do not have a result for one of these labs in the prior 30 days

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in Frequency of Hemoglobin A1c (A1c) and Thyroid-Stimulating Hormone (TSH) Ordered within 30 days of Prior Results | Study month 6
  This measure evaluates the impact of a randomized Our Practice Advisory (OPA) intervention on the frequency of Hemoglobin A1c (A1c) and Thyroid-Stimulating Hormone (TSH) tests ordered within 30 days of prior results. Data will be extracted from the UCLA Health Electronic Health Record (EHR) system using a structured query to identify qualifying test orders. Logistic regression will be used to compare the likelihood of A1c or TSH orders within the 30 days between the intervention and control group, adjusting for patient age, sex, and comorbidities. Clustering by providers will be accounted for.

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Health System, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No